CLINICAL TRIAL: NCT07016685
Title: Prognostic Factors for 90-day Mortality in Patients Undergoing Veno-venous Extracorporeal Membrane Oxygenation for Emergency Thoracic Surgery
Brief Title: Prognosis of Veno-Venous Extracorporeal Membrane Oxygenation in Emergency Thoracic Surgery
Acronym: PECUR
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: PI2025_843_0071
Record Dates: First submitted 2025-04-29; First posted 2025-06-12 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: VV-ECMO; Thoracic Surgery; Emergency Surgery; ARDS; Retrospective Cohort; Propensity Score Matching; Mortality; ECMO Outcomes
Keywords: thoracic surgery; VV-ECMO; emergency surgery; ARDS; retrospective cohort; propensity score matching; mortality; ECMO outcomes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VV-ECMO after emergency thoracic surgery: VV-ECMO after emergency thoracic surgery
- VV-ECMO for medical ARF: VV-ECMO for medical indication

SUMMARY:
Veno-vneous extracorporeal membrane oxygenation (VV-ECMO) is an established support strategy for acute respiratory failure, but its role in the perioperative management of emergency thoracic surgery remains poorly defined. This retrospective, multicenter, observational study aims to assess the clinical outcomes and prognostic factors in this high-risk population. Patients undergoing emergency thoracic procedures requiring VV-ECMO will be compared to a control cohort of patients treated with VV-ECMO for medical respiratory failure. Data will be collected from two French academic centers (CHU Amiens-Picardie and CHU Dijon).

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years
* VV-ECMO initiated during or after emergency thoracic surgery
* No opposition to data use

Exclusion Criteria:

* Pregnant women
* Veno-Arterial ECMO patients
* Patients under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults ≥ 18 years, Patients undergoing emergency thoracic procedures requiring VV-ECMO and patients treated with VV-ECMO for medical respiratory failure.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
90-day all-cause mortality | 90 days

SECONDARY OUTCOMES:
90-day mortality in oncologic vs. non-oncologic thoracic surgery | 90 days
Postoperative complication rates | 90 days
  Postoperative complication rates (hemorrhagic, thrombotic, infectious)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beyls C, Soulier-Zaninka Q, Georges O, Nguyen M, Dheilly T, Nicolas M, Huette P, De Dominicis F, Abou-Arab O, Guinot PG, Mahjoub Y. Perioperative Veno-Venous Extracorporeal Membrane Oxygenation in Non-Elective Thoracic Surgery: A Propensity-Matched Bicentric Comparison With Medical Indication. Interdiscip Cardiovasc Thorac Surg. 2025 Nov 6;40(11):ivaf255. doi: 10.1093/icvts/ivaf255. PMID 41134639